CLINICAL TRIAL: NCT05094388
Title: Validation of Prediction Model of Vitamin D Deficiency in Critically Ill Patients
Brief Title: Validation of Prediction Model of Vitamin D Deficiency
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202106128RIND
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Critical Illness
Keywords: critical care; vitamin D
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients: Patients admitted to intensive care units
  Interventions: Other: Admitted to intensive care units

INTERVENTIONS:
Other: Admitted to intensive care units — Admitted to intensive care units

SUMMARY:
Many studies have pointed out that patients with vitamin D deficiency have a longer stay in the intensive care unit and a poor prognosis. The investigators' previous multi-center prospective observational study in Taiwan reveals that the prevalence of vitamin D deficiency in critically ill patients in northern Taiwan is 59%, and the prevalence of severe vitamin D deficiency is 18%. The investigators used the data of that observational study to train a predictive model for predicting vitamin D deficiency. In addition, the association between vitamin D and the immune regulation of critically ill patients in Taiwan has not been investigated. This study aims primarily to validate the performance of the prediction model of vitamin D deficiency. Moreover, this study will investigate the association between vitamin D level and inflammatory cytokine levels.

This multi-center prospective observational study will enroll critically ill patients admitted to intensive care units (ICUs) less than 28 days. After inform consent, blood will be drawn for examination of vitamin D, interleukin 6, and interleukin 10 levels. The main diagnosis of ICU admission, past medical history, vital signs within 24 hours of admission, disease severity, and laboratory data will be recorded. The predictive model will use the required parameters to predict the patient's risk of vitamin D deficiency and vitamin D severe deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to intensive care units

Exclusion Criteria:

* aged < 20 years
* admitted to intensive care unit longer than 28 days
* body max index < 18 kg/m2
* receive vitamin D supplement > 3000 IU/day
* previously admitted to intensive care unit within 3 months
* have parathyroid disease, rickets, or severe liver cirrhosis [Child C]

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic | 1 day
  Area under the receiver operating characteristic of the prediction model of vitamin D deficiency

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No